CLINICAL TRIAL: NCT04212221
Title: A Multicenter, Open-label, Phase I/II Dose Escalation and Expansion Clinical Study to Assess the Safety and Efficacy of MGD013 Monotherapy and in Combination With Brivanib Alaninate (ZL-2301) in Patients With Advanced Liver Cancer
Brief Title: MGD013 Monotherapy and Combination With Brivanib Dose Escalation and Expansion Study in Advanced Liver Cancer Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to the rapid shifting of liver cancer disease landscape and the company's adjustment of development strategy.
Sponsor: Zai Lab (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Zai Lab (Hong Kong), Ltd. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZL-MGD013-202
Record Dates: First submitted 2019-12-19; First posted 2019-12-26 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-06

CONDITIONS: Advanced Hepatocellular Carcinoma (HCC)
MeSH Terms: interventions — brivanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MGD013 (Experimental): MGD013 monotherapy dose escalation and expansion
  Interventions: Drug: MGD013 monotherapy
- MGD013+Brivanib Alaninate (Experimental): MGD013+Brivanib Alaninate dose escalation and expansion
  Interventions: Drug: MGD013 in combination with Brivanib Alaninate

INTERVENTIONS:
Drug: MGD013 monotherapy — MGD013 monotherapy will start from Phase I dose escalation first, starting dose will be 120mg Q2W, the dose level may escalate sequentially following traditional 3+3 dose escalation scheme (120mg, 240mg, 400mg, 600mg) to determine the RP2D(recommended phase II dose) of MGD013 monotherapy. Then Phase II dose expansion study will initiate, patients will receive the fixed dose of MGD013 monotherapy with RP2D determined in Phase I study.
  Arms: MGD013
Drug: MGD013 in combination with Brivanib Alaninate — After determining the RP2D of MGD013 monotherapy, MGD013 at the fixed dose will be combined with Brivanib Alaninate. Dose escalation study of the combination therapy in Phase I will adopt traditional 3+3 dose escalation scheme; the dosage of Brivanib will start from 200 mg QD, and may escalate to 400 mg QD, 600 mg QD and a maximum of 800 mg QD to to determine the RP2D of MGD013 in combination with Brivanib Alaninate. Then Phase II dose expansion study will initiate, patients will receive the fixed dose of MGD013 and Brivanib Alaninate combination therapy with RP2D determined in Phase I study.
  Arms: MGD013+Brivanib Alaninate

SUMMARY:
This study consists of two parts: Phase I is a dose escalation study to determine the Recommended Phase II Dose (RP2D) of MGD013 monotherapy and that of MGD013 when in combination with Brivanib Alaninate (ZL-2301) in subjects with advanced liver cancer (including hepatocellular carcinoma and intrahepatic cholangiocarcinoma). Phase II is a dose expansion study and consists of two parts: Part 1 is to assess the safety and efficacy of MGD013 monotherapy and MGD013 in combination with ZL-2301 in subjects with advanced hepatocellular carcinoma (HCC); in Part 2, a therapeutic method (MGD013 monotherapy or MGD013 in combination with ZL-2301, determined by the sponsor according to the obtained data) will be selected for dose expansion study in HCC subjects who have previously failed immune checkpoint inhibitor treatment, to further evaluate the safety and efficacy of the study treatments in the specific group of subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who voluntarily sign the informed consent form (ICF);
2. Male or female subjects who are aged 18-75 years old;
3. Subjects with histologic, cytologic or clinical confirmed diagnosis of advanced HCC (Phase I could include intrahepatic cholangiocarcinoma or mixed hepatocellular-cholangiocarcinoma), and are not suitable for surgery or loco-regional therapy or have progressed following surgery and/or loco-regional therapy;
4. Subject who has at least one measurable lesion according to RECIST v1.1 criteria.
5. Phase I study: subjects who have previously received at least one line of systemic therapy, including immune checkpoint inhibitors, molecular targeted drugs or systematic chemotherapy, alone or in combination, and failed (progression confirmed by imaging) or were intolerant at the discretion of investigator; PhaseII：Advanced HCC cohort with subjects who have previously received immune checkpoint inhibitor treatment: subjects who have failed (progression confirmed by imaging) prior one line immune checkpoint inhibitor treatment, including anti-PD-1 antibody/anti-PD-L1 antibody and / or anti-CTLA-4 antibody, and/or molecular targeted therapy or systematic chemotherapy (monotherapy or in combination); Phase II: Advanced HCC cohort with subjects who have not previously received immune checkpoint inhibitor treatment: subjects who have failed (progression confirmed by imaging) or were intolerant to (at the discretion of investigator) previous molecular targeted therapy or systematic chemotherapy, without receiving immune checkpoint inhibitor treatment (including anti-PD-1 antibody, anti-PD-L1 antibody, anti-CTLA-4 antibody, and bispecific antibodies including the above targets).
6. Previous anti-tumor therapy must be completed no less than 2 weeks prior to the study treatment and all adverse events related to previous treatment must have recovered to CTCAE Grade ≤1; if subjects who have received prior immune checkpoint inhibitors have immune-related endocrinopathy, it should be controlled with hormone replacement therapy.
7. Phase I: Child-Pugh Class A; Phase II: Child-Pugh Class A or B with a score of ≤ 7;
8. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1;
9. Subjects with life expectancy ≥12 weeks;
10. Subjects with chronic HBV infection must have HBV-DNA <500 IU/ml, and have received at least 14 days of anti-HBV treatment (e.g. entecavir, tenofovir) prior to the initiation of study treatment and are willing to receive antiviral treatment throughout the study; Subjects with RNA-positive HCV must have received standard antiviral treatment and the elevation of their liver enzymes must not exceed the level of CTCAE Grade 1;
11. Adequate vital organ function as shown below:

(1) Blood system function (subjects must have not received blood transfusion or stimulating growth factors within 14 days prior to screening test): neutrophil count ≥1.5×109/L, platelet count ≥ 75×109/L, hemoglobin ≥ 90 g/L; (2) Liver and kidney function (no albumin transfusion within 14 days prior to screening test): serum total bilirubin ≤ 2.5×ULN, serum albumin ≥ 29 g/L, ALT and AST ≤ 5×ULN; serum creatinine <1.5×ULN or eGFR (Cockcroft-Gault formula) ≥ 60 ml/min; (3) Coagulation function: international normalized ratio (INR)≤2.3 or prothrombin time (PT) of ≤ 6 seconds above control; (4) Left ventricular ejection fraction (LVEF) ≥50% by two-dimensional echocardiography.

12. Female subjects (except for females who have underwent surgical sterilization and those have been menopausal for more than one year) who are of childbearing potential are required to adopt a medically proven method for contraception (e.g. intrauterine contraception device, contraceptive pill or condom) throughout the study and up to 120 days after the last dose of investigational products; females who are of childbearing age and who do not underwent surgical sterilization must have negative serum or urine HCG tests within 7 days prior to enrollment; female subjects must not be breastfeeding; male subjects whose partners are of childbearing potential should use effective contraceptive methods throughout the study and up to 120 days after the last dose of investigational product.

13. Subjects who are willing to provide oncological tissues (if applicable) for biomarker test.

Exclusion Criteria:

1. Subjects who have known fibrolamellar carcinoma of liver for phase I and subjects who have fibrolamellar carcinoma, mixed HCC- cholangiocarcinoma or cholangiocarcinoma for phase II;
2. Subjects with brain metastasis or leptomeningeal metastasis confirmed by brain MRI during screening period;
3. Subjects with a diagnosis of other malignant tumors within 5 years prior to first administration, except for skin basal cell carcinoma, skin squamous cell carcinoma and/or in situ cancer following radical resection;
4. Subjects who had liver or other sites loco-regional treatment (including transcatheter arterial chemoembolization (TACE), transcatheter arterial embolization (TAE), hepatic artery infusion (HAI), local radiotherapy, radioembolization, radiofrequency ablation, cryoablation or percutaneous ethanol injection) , or who had major surgery of liver or other sites within 4 weeks prior to first administration, or had minor surgical procedures (e.g. simple excision, tooth extraction) within one week prior to first administration, or had received palliative radiotherapy for bone metastasis within 2 weeks and radiotherapy-related toxicity ≥ CTCAE Grade 2.
5. Subjects who have moderate or severe ascites (detected by B-ultrasound or CT), or require therapeutic abdominal paracentesis or drainage;
6. Subjects with a history of hepatic encephalopathy;
7. Subjects with a history of unhealed wounds or ulcers or bone fractures within 3 months prior to study enrollment;
8. Subjects who plan to have or had allogenic organ or bone marrow transplantation;
9. Subjects who are at increased risk of bleeding or have history of thrombosis:

(1) Clinically significant bleeding within 3 months prior to screening or clear bleeding tendency; (2) Gastrointestinal hemorrhage within 6 months prior to screening or clear tendency of gastrointestinal hemorrhage; (3) Arterial/venous thromboembolic events within 6 months prior to screening, such as cerebrovascular accident (including transient ischemic attack), pulmonary embolism, etc.; (4) Require anticoagulation therapy with an agent such as warfarin or heparin; (5) Require chronic anti-platelet therapy (such as aspirin≥100 mg/day, clopidogrel, etc.); 10. Subjects who have clinically significant cardiovascular diseases:

1. NYHA (New York Heart Association)stage 3 and 4 congestive heart failure;
2. Unstable angina pectoris or newly diagnosed angina pectoris or myocardial infarction within 12 months prior to screening;
3. Arrhythmias requiring medications other than β-blockers;
4. Valvular heart disease of ≥ CTCAE grade 2;
5. Hypertension inadequately controlled by drugs (systolic pressure >150 mmHg or diastolic pressure >90 mmHg); 11. Subjects who have history of symptomatic pulmonary fibrosis, or have interstitial pneumonitis, pneumoconiosis, radiation pneumonitis, drug-related pneumonitis, severe impairment of pulmonary function, or other suspicious pulmonary diseases that may interfere with drug-related pulmonary toxicity detection and treatment; 12. Subjects who have suffered active bacterial or fungal infections requiring systemic treatment within 7 days prior to screening; or active tuberculosis; 13. Subjects with active co-infection of Hepatitis B and C, confirmed by positive HBV surface antigen or HBV DNA and HCV RNA 14. Subjects who have any active, known or suspected autoimmune disease; 15. Subjects with a condition requiring systematic treatment with corticosteroids (>10 mg/day prednisone or equivalent) or other immunosuppressive drugs within 14 days before administration of the investigational drug. In the absence of active autoimmune diseases, inhalation or topical use of steroids (>10 mg/day prednisone or equivalent) is allowed; 16. Other laboratory abnormalities:

(1) Hyponatremia, hypokalemia or hypophosphatemia that have occurred before the first administration, and failed to restore to normal level after electrolyte supplementation therapy; (2) Confirmed diagnosis of thyroid dysfunction, which cannot be maintained within normal range following thyroid hormone replacement therapy; (3) Positive Human immunodeficiency virus (HIV) test; 17. QTc interval >480 ms on two consecutive ECGs; 18. Female subjects during pregnancy or lactation; female subjects of childbearing potential or male subjects who are not willing to use contraception or contraceptive measures during the study; 19. Subjects who have previously received two lines and above tumor immune checkpiont inhibitor treatment, mainly including anti-PD-1, anti-PD-L1 and anti-CTLA-4 antibodies, etc, or bispecific antibodies including the above targets, or received anti-LAG-3 antibody; whether subjects who have previously received other tumor immunotherapy can be enrolled should be determined by the sponsor; 20. Known or suspected history of severe allergy to investigational drugs; 21. Subjects who have received live attenuated vaccines or any investigational drugs that have not been marketed in China within 4 weeks prior to first administration; 22. If subjects who have previously used immune checkpoint inhibitors (such as anti-PD-1, anti-PD-L1, anti-CTLA-4 antibodies) have the following drug-related adverse events, they will be not suitable for inclusion regardless of recovered or not:

1. ≥ Grade 3 eye-related adverse events
2. Grade 4 abnormal liver function
3. ≥ Grade 3 neurotoxicity
4. ≥ Grade 3 colitis
5. ≥ Grade 3 renal toxicity
6. ≥ Grade 3 pneumonitis 23. Subjects who are not suitable for inclusion as judged by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ZhengGang Ren, PhD, Principal Investigator — Fudan University
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consists of two phases: Phase I dose escalation and Phase II dose expansion. A total of 89 participants were enrolled in the study across 16 centers in China, including 82 participants who received at least one dose of MGD013 and 7 participants who received at least one dose of MGD013 in combination with Brivanib alaninate.
Groups:
- Phase 1: MGD013 120mg: Participants received 120 mg MGD013 intravenously once every 2 weeks (Q2W).
- Phase 1: MGD013 240mg: Participants received 240 mg MGD013 intravenously once every 2 weeks (Q2W).
- Phase 1: MGD013 400mg: Participants received 400 mg MGD013 intravenously once every 2 weeks (Q2W).
- Phase 1: MGD013 600mg: Participants received 600 mg MGD013 intravenously once every 2 weeks (Q2W).
- Phase 1: MGD013 400mg + Brivanib 400mg: Participants received 400 mg MGD013 intravenously once every 2 weeks (Q2W), in combination with 400 mg Brivanib alaninate orally once daily (QD).
- Phase 1: MGD013 600mg + Brivanib 400mg: Participants received 600 mg MGD013 intravenously once every 2 weeks (Q2W), in combination with 400 mg Brivanib alaninate orally once daily (QD).
- Phase 2: MGD013 600mg Post-CPI Cohort: Participants who had received at least one prior line of systemic therapy including prior immune checkpoint inhibitor (CPI) treatment received 600 mg MGD013 intravenously once every 2 weeks (Q2W).
- Phase 2: MGD013 600mg CPI-naive Cohort: Participants who had received at least one prior line of systemic therapy without prior immune checkpoint inhibitor (CPI) treatment received 600 mg MGD013 intravenously once every 2 weeks (Q2W).
Period: Overall Study
Arm/Group | Phase 1: MGD013 120mg | Phase 1: MGD013 240mg | Phase 1: MGD013 400mg | Phase 1: MGD013 600mg | Phase 1: MGD013 400mg + Brivanib 400mg | Phase 1: MGD013 600mg + Brivanib 400mg | Phase 2: MGD013 600mg Post-CPI Cohort | Phase 2: MGD013 600mg CPI-naive Cohort
Started | 1 | 3 | 3 | 6 | 3 | 4 | 33 | 36
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 3 | 3 | 6 | 3 | 4 | 33 | 36
Not completed — Remained on Treatment | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 9
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Disease progression according to irRECIST | 1 | 2 | 3 | 3 | 2 | 2 | 21 | 17
Not completed — Global Deterioration of Health Status | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Investigator's Decision | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0
Not completed — Participant refused to continue treatment | 0 | 1 | 0 | 1 | 1 | 2 | 4 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All patients who received at least one dose of study treatment (any component of combination treatment whichever is first).
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: MGD013 120mg | Phase 1: MGD013 240mg | Phase 1: MGD013 400mg | Phase 1: MGD013 600mg | Phase 1: MGD013 400mg + Brivanib 400mg | Phase 1: MGD013 600mg + Brivanib 400mg | Phase 2: MGD013 600mg Post-CPI Cohort | Phase 2: MGD013 600mg CPI-naive Cohort | Total
Number analyzed (Participants) | 1 | 3 | 3 | 6 | 3 | 4 | 33 | 36 | 89
Age, Customized [Count of Participants; unit: Participants]
  Age Group: < 65 Years | 0 | 0 | 2 | 3 | 0 | 3 | 26 | 26 | 60
  Age Group: ≥ 65 Years | 1 | 3 | 1 | 3 | 3 | 1 | 7 | 10 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 2 | 10
  Male | 1 | 3 | 3 | 6 | 3 | 3 | 26 | 34 | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 3 | 3 | 6 | 3 | 4 | 33 | 36 | 89
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: DLT was defined as the adverse events (AEs) listed in the protocol occurring within 4 weeks (the first 2 cycles, 28 days) after the investigational drugs which were at least possibly related to the study drugs. AE severity was graded from 1 to 5 according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0.
Time Frame: The first two cycles (Cycle 1 and Cycle 2) of the study treatment(s). A cycle lasted for two weeks (14 days) in the study.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: MGD013 120mg | Phase 1: MGD013 240mg | Phase 1: MGD013 400mg | Phase 1: MGD013 600mg | Phase 1: MGD013 400mg + Brivanib 400mg | Phase 1: MGD013 600mg + Brivanib 400mg
Number analyzed (Participants) | 1 | 3 | 3 | 6 | 3 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Phase 1 and Phase 2: Safety
Description: All adverse events (AEs) occurring on or after the first study treatment were listed and summarized. Treatment-Emergent Adverse Event (TEAE) was defined as an AE that had an onset date or a worsening in severity from baseline on or after the first dose of study treatment (any component of combination treatment whichever is first) up to 30 days following study treatment (any component of combination treatment whichever was last) discontinuation. All adverse events were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0.
Time Frame: AEs would be collected throughout the clinical trial, from the signing of the informed consent form (ICF) to the end of the trial (until 30 days after the last dose of investigational drugs). Up to approximately 24 months.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: MGD013 120mg | Phase 1: MGD013 240mg | Phase 1: MGD013 400mg | Phase 1: MGD013 600mg | Phase 1: MGD013 400mg + Brivanib 400mg | Phase 1: MGD013 600mg + Brivanib 400mg | Phase 2: MGD013 600mg Post-CPI Cohort | Phase 2: MGD013 600mg CPI-naive Cohort
Number analyzed (Participants) | 1 | 3 | 3 | 6 | 3 | 4 | 33 | 36
Participants
  Patients with at Least One TEAE | 1 | 3 | 3 | 6 | 3 | 4 | 31 | 34
  TEAEs with Grade 3 or Higher | 1 | 1 | 0 | 2 | 1 | 2 | 11 | 10
  Serious TEAEs | 0 | 1 | 0 | 1 | 0 | 1 | 10 | 8
  TEAEs Leading to Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  TEAEs Leading to Treatment Discontinuation of Any Treatment Component | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
  TEAEs Leading to Dose Modification of Any Treatment Component | 1 | 2 | 0 | 1 | 2 | 3 | 13 | 15
  Treatment-Related TEAEs | 1 | 2 | 3 | 6 | 3 | 4 | 23 | 27
  Treatment-Related TEAEs with Grade 3 or Higher | 1 | 1 | 0 | 1 | 1 | 1 | 5 | 8
  Treatment-Related Serious TEAEs | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 6
  Treatment-Related TEAEs Leading to Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Treatment-Related TEAEs Leading to Treatment Discontinuation of Any Treatment Component | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
  Treatment-Related TEAEs Leading to Dose Modification of Any Treatment Component | 1 | 1 | 0 | 1 | 2 | 3 | 7 | 12

3. Primary Outcome: Phase 2: Objective Response Rate (ORR) Assessed by Blinded Independent Central Review (BICR) According to RECIST 1.1
Description: ORR was defined as the proportion of participants with a confirmed objective response, either complete response (CR) or partial response (PR), before progression based on RECIST v1.1. Participants who had no measurable disease at baseline and/or no post-baseline tumor assessment due to any reason will be considered nonresponders. An estimate of ORR was calculated for each treatment arm, and its 95% CI was calculated using the Clopper-Pearson method.
Time Frame: Radiologic examinations were conducted at baseline within 28 days prior to the start of study medication and every 8 weeks (±7 days) dated from the first day of the first cycle until disease progression. Up to approximately 24 months.
Population: All patients who received at least one dose of study treatment (any component of combination treatment whichever is first) in phase 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: MGD013 600mg Post-CPI Cohort | Phase 2: MGD013 600mg CPI-naive Cohort
Number analyzed (Participants) | 33 | 36
percentage of participants | 3.0 [0.08 to 15.76] | 8.3 [1.75 to 22.47]

4. Secondary Outcome: Phase 2: Objective Response Rate (ORR) by Investigator Assessment According to RECIST 1.1
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: MGD013 600mg Post-CPI Cohort | Phase 2: MGD013 600mg CPI-naive Cohort
Number analyzed (Participants) | 33 | 36
percentage of participants | 3.0 [0.08 to 15.76] | 11.1 [3.11 to 26.06]

5. Secondary Outcome: Phase 2: Disease Control Rate (DCR) by BICR / Investigator Assessment According to RECIST 1.1
Description: DCR was defined as the percentage of participants who attained a best overall response status of CR, PR, and SD. If best overall response is SD, the SD should be stable SD, that is the date of SD should be at least 6 weeks after first dose. DCR was analyzed using the same methodology as specified for ORR.
Time Frame: Radiologic examinations were conducted at basline within 28 days prior to the start of study medication and every 8 weeks (±7 days) dated from the first day of the first cycle until disease progression. Up to approximately 24 months.
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: MGD013 600mg Post-CPI Cohort | Phase 2: MGD013 600mg CPI-naive Cohort
Number analyzed (Participants) | 33 | 36
percentage of participants
  DCR by BICR Assessment | 33.3 [17.96 to 51.83] | 30.6 [16.35 to 48.11]
  DCR by Investigator Assessment | 45.5 [28.11 to 63.65] | 38.9 [23.14 to 56.54]

6. Secondary Outcome: Phase 2: Time to Response (TTR) by Investigator Assessment According to RECIST 1.1
Description: TTR was defined as the time from the first dose date to the date of the earliest confirmed response assessed using RECIST V1.1. Only responders were included in the analysis.
Time Frame: as for outcome 3
Population: as for baseline characteristics
Measure: Median (Full Range); unit: months
Arm/Group | Phase 2: MGD013 600mg Post-CPI Cohort | Phase 2: MGD013 600mg CPI-naive Cohort
Number analyzed (Participants) | 1 | 4
months | 1.70 [1.7 to 1.7] | 1.80 [1.7 to 3.5]

7. Secondary Outcome: Phase 2: Duration of Response (DoR) by Investigator Assessment According to RECIST 1.1
Description: DoR was defined for subjects with a confirmed objective response as the time from the first occurrence of response (CR or PR) to disease progression or death, whichever occurred first. Participants who had no progression or death would be censored.
Time Frame: as for outcome 3
Population: as for baseline characteristics
Measure: Median (Full Range); unit: months
Arm/Group | Phase 2: MGD013 600mg Post-CPI Cohort | Phase 2: MGD013 600mg CPI-naive Cohort
Number analyzed (Participants) | 1 | 4
months | 9.20 [9.2 to 9.2] | 5.80 [3.7 to 5.8]

8. Secondary Outcome: Phase 2: Progression-Free Survival (PFS) by Investigator Assessment According to RECIST 1.1
Description: PFS was defined as the time from the date of first dose of study treatment (any component of combination treatment whichever is first) to the first documented disease progression as determined by the investigator or BICR with the use of RECIST v1.1, or death from any cause, whichever occurred first. Kaplan-Meier methodology was used to estimate the median PFS for each treatment arm and to construct survival curves for each treatment arm. The Brookmeyer-Crowley methodology was used to construct the 95% CI for the median PFS for each treatment arm (Brookmeyer and Crowley 1982).
Time Frame: as for outcome 3
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: MGD013 600mg Post-CPI Cohort | Phase 2: MGD013 600mg CPI-naive Cohort
Number analyzed (Participants) | 33 | 36
months | 2.40 [1.90 to 4.10] | 3.05 [1.90 to 5.60]

9. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS was defined as the time from the date of the first dose of study treatment (any component of combination treatment whichever was first) to the date of death from any cause. Participants who were alive at the time of the analysis data cutoff would be censored at the last date they were known to be alive. Participants with no post-baseline information were censored at the date of the first dose of study treatment (any study treatment component for combo therapy).
Time Frame: From the date of the first dose of study treatment to the date of death from any cause. Up to approximately 24 months.
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: MGD013 600mg Post-CPI Cohort | Phase 2: MGD013 600mg CPI-naive Cohort
Number analyzed (Participants) | 33 | 36
months | NA [9.70 to NA] — The median and the upper bound of the confidence interval could not be estimated because of insufficient number of events. | NA [7.10 to NA] — The median and the upper bound of the confidence interval could not be estimated because of insufficient number of events.

10. Secondary Outcome: Phase 1: Objective Response Rate (ORR) by Investigator Assessment According to RECIST 1.1
Description: as for outcome 3
Time Frame: as for outcome 3
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: MGD013 120mg | Phase 1: MGD013 240mg | Phase 1: MGD013 400mg | Phase 1: MGD013 600mg | Phase 1: MGD013 400mg + Brivanib 400mg | Phase 1: MGD013 600mg + Brivanib 400mg
Number analyzed (Participants) | 1 | 3 | 3 | 6 | 3 | 4
percentage of participants | 0 [0.00 to 97.50] | 33.3 [0.84 to 90.57] | 0 [0.00 to 70.76] | 16.7 [0.42 to 64.12] | 0 [0.00 to 70.76] | 0 [0.00 to 60.24]

11. Secondary Outcome: Phase 1: Disease Control Rate (DCR) by Investigator Assessment According to RECIST 1.1
Description: as for outcome 5
Time Frame: as for outcome 5
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: MGD013 120mg | Phase 1: MGD013 240mg | Phase 1: MGD013 400mg | Phase 1: MGD013 600mg | Phase 1: MGD013 400mg + Brivanib 400mg | Phase 1: MGD013 600mg + Brivanib 400mg
Number analyzed (Participants) | 1 | 3 | 3 | 6 | 3 | 4
percentage of participants | 100 [2.50 to 100.0] | 100 [29.24 to 100.0] | 33.3 [0.84 to 90.57] | 16.7 [0.42 to 64.12] | 0 [0.00 to 70.76] | 25.0 [0.63 to 80.59]

ADVERSE EVENTS:
Time Frame: From the date of administration of the first dose of study treatment (any component of combination treatment whichever is first) up to 30 days following study treatment discontinuation (any component of combination treatment whichever is last). Adverse event reporting for all-cause mortality considers all deaths that occurred during the study. Up to approximately 24 months.
Arm/Group | Phase 1: MGD013 120mg | Phase 1: MGD013 240mg | Phase 1: MGD013 400mg | Phase 1: MGD013 600mg | Phase 1: MGD013 400mg + Brivanib 400mg | Phase 1: MGD013 600mg + Brivanib 400mg | Phase 2: MGD013 600mg Post-CPI Cohort | Phase 2: MGD013 600mg CPI-naive Cohort
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/3 | 0/3 | 1/6 | 2/3 | 1/4 | 10/33 | 11/36
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/3 | 0/3 | 1/6 | 0/3 | 1/4 | 10/33 | 8/36
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3 | 3/3 | 6/6 | 3/3 | 4/4 | 30/33 | 34/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: MGD013 120mg (N=1) | Phase 1: MGD013 240mg (N=3) | Phase 1: MGD013 400mg (N=3) | Phase 1: MGD013 600mg (N=6) | Phase 1: MGD013 400mg + Brivanib 400mg (N=3) | Phase 1: MGD013 600mg + Brivanib 400mg (N=4) | Phase 2: MGD013 600mg Post-CPI Cohort (N=33) | Phase 2: MGD013 600mg CPI-naive Cohort (N=36)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: MGD013 120mg (N=1) | Phase 1: MGD013 240mg (N=3) | Phase 1: MGD013 400mg (N=3) | Phase 1: MGD013 600mg (N=6) | Phase 1: MGD013 400mg + Brivanib 400mg (N=3) | Phase 1: MGD013 600mg + Brivanib 400mg (N=4) | Phase 2: MGD013 600mg Post-CPI Cohort (N=33) | Phase 2: MGD013 600mg CPI-naive Cohort (N=36)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 3 | 7
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 5
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 4
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 5
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 5
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4
Asthenia (General disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 3 | 3
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 5
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 2 | 2 | 1 | 6 | 3
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1
Tongue injury (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 1 | 2 | 1 | 1 | 4 | 11
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 4 | 0 | 1 | 7 | 9
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 4 | 2 | 0 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 3 | 0 | 0 | 4 | 10
Blood bilirubin unconjugated increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Free fatty acids increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Hepatitis B DNA increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 3
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 4
Platelet count decreased (Investigations) | 0 | 0 | 2 | 2 | 1 | 1 | 7 | 8
Protein urine present (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Prothrombin level decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Total bile acids increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Tri-iodothyronine decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tri-iodothyronine free decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urine ketone body present (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 4 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 3
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 3 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4 | 2 | 2 | 5 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 7 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 2 | 1 | 1 | 8 | 5
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inadequate diet (Social circumstances) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/21/NCT04212221/Prot_SAP_000.pdf